CLINICAL TRIAL: NCT03430609
Title: Ovarian Function After Use of Various Hemostatic Techniques During Treatment for Endometrioma: A Randomized Control Trial
Brief Title: Ovarian Function After Use of Various Hemostatic Techniques During Treatment for Endometrioma
Acronym: Endometrioma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Collaborators: Federal University of Paraíba (Other); Irmandade da Santa Casa de Misericordia de Sao Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1203-2508; 71621717.9.0000.8069 (Other: Certificate of Presentation for Ethical Assessment (CAAE))
Record Dates: First submitted 2017-10-31; First posted 2018-02-13 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Endometriosis Ovary; Laparoscopy; Ovary; Functional Disturbance; Hemostasis
Keywords: endometrioma; laparoscopy; ovarian reserve; anti-mullerian hormone
MeSH Terms: conditions — Endometriosis | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Open-label randomized clinical trial to be conducted at Lauro Wanderley University Hospital, at Federal University of Paraiba, from September 2017 to August 2020. Eighty-four patients will be randomly allocated to three groups according to the hemostatic technique used during laparoscopic surgery for ovarian endometrioma: bipolar coagulation, laparoscopic suture and hemostatic matrix. Ovarian function will be assessed by measuring serum anti-Mullerian hormone and by ultrasound antral follicle counts before surgery and 1, 3 and 6 months after surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Bipolar tweezers Astus Medical© (Active Comparator): Laparoscopic treatment for endometrioma Astus© will use Bipolar coagulation (bipolar tweezers, Astus Medical ©, Copyright 2015, Tampa FL, USA) with 30 W power and a Valleylab generator (Medronic ©, Copyright 2017, Medtronic Parkway, Minneapolis, USA); the number of coagulated points will be counted, and the time for coagulation will be measured in seconds. Transvaginal ultrasound for antral follicle count and blood collection will be performed in this group of patients before surgery, 1, 3 and 6 months after the procedure to dose AMH level, FSH level and to count the number of antral follicle.
  Interventions: Procedure: Laparoscopic treatment for endometrioma Astus©; Diagnostic Test: AMH Level; Diagnostic Test: Transvaginal ultrasound for antral follicle count
- 2-0 Vicryl® Suture (Active Comparator): Laparoscopic treatment for endometrioma Vicryl® will use suturing with simple suture (2-0/Vicryl polyglactin absorbable synthetic suture; Ethicon Inc., New Jersey, USA); the number of sutures will be recorded. Transvaginal ultrasound for antral follicle count and blood collection will be performed in this group of patients before surgery, 1, 3 and 6 months after the procedure to dose AMH level, FSH level and to count the number of antral follicle.
  Interventions: Diagnostic Test: AMH Level; Diagnostic Test: Transvaginal ultrasound for antral follicle count; Procedure: Laparoscopic treatment for endometrioma Vicryl®
- Surgicel® (Active Comparator): Laparoscopic treatment for endometrioma Surgicel® will use Hemostatic matrix (Surgicel® Original Absorbable Hemostat, Ethicon, USA). Transvaginal ultrasound for antral follicle count and blood collection will be performed in this group of patients before surgery, 1, 3 and 6 months after the procedure to dose AMH level, FSH level and to count the number of antral follicle.
  Interventions: Diagnostic Test: AMH Level; Diagnostic Test: Transvaginal ultrasound for antral follicle count; Procedure: Laparoscopic treatment for endometrioma Surgicel®

INTERVENTIONS:
Procedure: Laparoscopic treatment for endometrioma Astus© — Laparoscopic surgery will be performed by the same surgeon, according to the routine of the service.In all of the groups, endometrioma will be removed by means of the traction and countertraction techniques. Adhesiolysis will be performed to separate the ovary from the adjacent structures as needed. In case of cyst rupture, the contents will be aspirated, and the site where the endometrioma contents fell will be exhaustively rinsed. In the hemostasis , the investigators will use coagulation with bipolar tweezers Astus Medical© in this group.
  Other Names: Treatment for ovarian endometrioma with bipolar Astus©
  Arms: Bipolar tweezers Astus Medical©
Diagnostic Test: AMH Level — The AMH levels will be quantitatively measured via ELISA, Enzyme-Linked Immunosorbent Assay (Diagnostic Systems Laboratories, Webster, TX), with a detection sensitivity of 0.006 ng/mL.
  The participants' sera will be obtained from blood samples after centrifugation for 10 minutes to separate the cell contents and debris. Each serum sample will be transferred to polypropylene tubes and stored at -70ºC. Venous blood samples will be collected before surgery (on the day ultrasound is performed for antral follicle count, approximately 1 month before surgery) and 1, 3 and 6 months after surgery.
  Other Names: Antimulerian Hormone
Diagnostic Test: Transvaginal ultrasound for antral follicle count — The participants will be subjected to transvaginal ultrasound for antral follicle count before surgery (1 month before surgery) and 1, 3 and 6 months after surgery. This test will be performed during the early proliferative stage (days 3 to 6 of the menstrual cycle); the size of the endometrioma and the ovary volume will be recorded, and functional cysts or suspected malignant cysts will be ruled out. For measurement of cysts, the average diameter of the three perpendicular ovary dimensions will be considered. For antral follicle count, the total number of follicles with diameters under 9 mm will be considered.
  Other Names: AFC
Procedure: Laparoscopic treatment for endometrioma Vicryl® — Laparoscopic surgery will be performed by the same surgeon, according to the routine of the service.In all of the groups, endometrioma will be removed by means of the traction and countertraction techniques. Adhesiolysis will be performed to separate the ovary from the adjacent structures as needed. In case of cyst rupture, the contents will be aspirated, and the site where the endometrioma contents fell will be exhaustively rinsed. In the hemostasis , the investigators will perform suture with 2-0 Vicryl® in this group.
  Other Names: Treatment for ovarian endometrioma using vicryl suture
  Arms: 2-0 Vicryl® Suture
Procedure: Laparoscopic treatment for endometrioma Surgicel® — Laparoscopic surgery will be performed by the same surgeon, according to the routine of the service.In all of the groups, endometrioma will be removed by means of the traction and countertraction techniques. Adhesiolysis will be performed to separate the ovary from the adjacent structures as needed. In case of cyst rupture, the contents will be aspirated, and the site where the endometrioma contents fell will be exhaustively rinsed. In this group, for hemostasis , the investigators will use matrix Surgicel®
  Other Names: Treatment for ovarian endometrioma using matrix Surgicel®
  Arms: Surgicel®

SUMMARY:
Background: Endometriosis is defined by the presence of endometrial tissue outside the uterine cavity due to causes not yet fully elucidated. The disease affects approximately 2% of women of reproductive age and is associated with infertility. Approximately 17% to 44% of women with endometriosis exhibit endometrioma, or ovarian endometriosis. Laparoscopic cystectomy is currently considered the gold standard treatment for this problem, resulting in improvement of symptoms, a lower recurrence rate and a higher pregnancy rate among infertile patients. However, several studies have shown that this treatment is not free from risks because it is associated with reduction of the ovarian reserve due to accidental removal of ovarian cortex during stripping of the capsule or damage caused by the coagulation energy during hemostasis, even when performed by experienced surgeons. There is still controversy in the literature as to the cause of the reduction of the ovarian reserve, as the mere presence of endometrioma reduces ovarian function by itself. The aim of this study is to compare the effects of different hemostatic methods on the ovarian function of women subjected to laparoscopic surgery for ovarian endometrioma.

Methods: Open-label randomized clinical trial to be conducted at Lauro Wanderley University Hospital from September 2017 to August 2020. Eighty-four patients will be randomly allocated to three groups according to the hemostatic technique used during laparoscopic surgery for ovarian endometrioma: bipolar coagulation, laparoscopic suture and hemostatic matrix. Ovarian function will be assessed by measuring serum anti-Mullerian hormone and follicle-stimulating hormone levels and by ultrasound antral follicle counts before surgery and 1, 3 and 6 months after surgery. The study was approved by the research ethics committee at the Medical Sciences Center, Federal University of Paraíba CAAE no. 71621717.9.0000.8069.

Discussion: The present study intends to assess the ovarian function of patients with endometrioma subjected to laparoscopic surgical treatment, comparing different hemostatic techniques like bipolar coagulation versus suture versus hemostatic matrix with objective assessments of bipolar coagulation to avoid bias. Thus, the investigators expect to contribute data likely to dispel doubts on the subject.

DETAILED DESCRIPTION:
OBJECTIVES

To compare the effects of various hemostatic methods on the ovarian function of patients subjected to laparoscopic surgery for ovarian endometrioma through AMH and ultrasound antral follicle count (AFC).

METHODS

Study design

An open-label randomized clinical trial will be performed to compare the impact of hemostatic techniques like bipolar coagulation versus laparoscopic suture versus hemostatic matrix during laparoscopic surgery for ovarian endometrioma on the ovarian follicular reserve.

Study setting

The study will be conducted at the endoscopic gynecology unit of Lauro Wanderley University Hospital, Federal University of Paraíba in Brazil.

Study and data collection period

The study will be performed from September 2017 to August 2020. Data will be collected from October 2017 to April 2020.

Study population

Patients with ovarian cysts suggestive of endometrioma on ultrasound cared for at the outpatient clinic of the HULW endoscopic gynecology unit during the study period.

Sample

In compliance with the eligibility criteria, consecutive convenience sampling will be performed among patients with ovarian cysts suggestive of endometrioma on ultrasound subjected to laparoscopic surgery and randomized to receive different hemostatic techniques during surgery: bipolar coagulation, laparoscopic suture or hemostatic matrix.

Sample size. The sample size was calculated through resources available on the Laboratory of Epidemiology and Statistics website of the Dante Pazzanese Institute. The calculation was based on data provided by Sönmezer et al. In this article, the investigators detected significant difference in the first month postoperative, with 2.72±1.49 AMH measurement among patients who receive hemostatic matrix versus 1.64±0.93 among patients who receive bipolar coagulation. Then the statistical assume that the 1.49 standard deviation for AMH measurement in the first month was significant and was the number that provide a greater sample size when compared with other values from that article. The difference to be detected is 1.08, which corresponds to the mean difference in AMH in the first month between the patients who receive hemostatic matrix and bipolar coagulation. On those grounds, and to achieve adequate statistical power 80%; p=0.05, each group should consist of 23 participants. Considering possible losses, the sample will be increased by 20%, corresponding to 28 participants per group and a total of 84 women.

Following inclusion, the participants will be randomized as described below. The sample will be divided into three groups according to the hemostatic technique used:

1. Bipolar coagulation (bipolar tweezers, Astus Medical ©, Copyright 2015, Tampa FL, USA) with 30 W power and a Valleylab generator Medronic ©, Copyright 2017, Medtronic Parkway, Minneapolis, USA; the number of coagulated points will be counted, and the time for coagulation will be measured in seconds.
2. Laparoscopic suturing with simple suture 2-0/Vicryl polyglactin absorbable synthetic suture; Ethicon Inc., New Jersey, USA; the number of sutures will be recorded.
3. Hemostatic matrix Surgicel® Original Absorbable Hemostat, Ethicon, USA.

Procedures for randomization. Randomization to receive the various hemostatic techniques bipolar coagulation, laparoscopic suture or hemostatic matrix during laparoscopic surgery for endometrioma will be performed based on a list of sequential numbers from 1 to 84 total number of participants to be randomized generated by a statistician using Random Allocation Software version 2.0 and the letters A, B and C; the statistician will be blinded as to their meaning.

Another individual not participating in the study will receive the list of random numbers prepared by the statistician and will attribute a letter to each technique bipolar coagulation, laparoscopic surgery and hemostatic matrix through the lottery method. Next, this same individual will prepare opaque envelopes numbered from 1 to 84, which will contain the group of allocation.

At the time of inclusion, each participant will be assigned a number corresponding to their order of entrance in the study. The envelope with the corresponding number will be opened by a nurse at the surgical theater at the time of hemostasis during surgery. Thus, allocation will remain concealed before surgery.

Procedures for assessment of the ovarian reserve. The ovarian reserve will be assessed through measurements of AMH levels and ultrasound antral follicle count. The AMH levels will be quantitatively measured via ELISA, Enzyme-Linked Immunosorbent Assay Diagnostic Systems Laboratories, Webster, TX, with a detection sensitivity of 0.006 ng/mL.

The participants' sera will be obtained from blood samples after centrifugation for 10 minutes to separate the cell contents and debris. Each serum sample will be transferred to polypropylene tubes and stored at -70ºC. Venous blood samples will be collected before surgery on the day ultrasound is performed for antral follicle count, approximately 1 month before surgery and 1, 3 and 6 months after surgery.

The participants will also be subjected to transvaginal ultrasound for antral follicle count before surgery 1 month before surgery and 1, 3 and 6 months after surgery. This test will be performed during the early proliferative stage days 3 to 6 of the menstrual cycle; the size of the endometrioma and the ovary volume will be recorded, and functional cysts or suspected malignant cysts will be ruled out. For measurement of cysts, the average diameter of the three perpendicular ovary dimensions will be considered. For antral follicle count, the total number of follicles with diameters under 9 mm will be considered. The ovary and cyst volumes will be calculated using the equation 4/3 x π x (d/2)3, where d is the average diameter. All ultrasound tests will be performed by the same operator using the same device.

Procedures for laparoscopic surgery. Surgery will be performed by the same surgeon, with the participants under general anesthesia and in a semi-lithotomy position. A 10-mm umbilical puncture will be performed for the camera after insufflation of the pneumoperitoneum; three additional 5-mm punctures will be performed on the right iliac fossa, left iliac fossa and suprapubic area for instruments. The intra-abdominal pressure will be kept at approximately 15 mmHg.

Endometriosis will be categorized according to the classification formulated by the American Society for Reproductive Medicine - ASRM. In all of the groups, endometrioma will be removed by means of the traction and countertraction techniques. Adhesiolysis will be performed to separate the ovary from the adjacent structures as needed. In case of cyst rupture, the contents will be aspirated, and the site where the endometrioma contents fell will be exhaustively rinsed.

In the group allocated to receive bipolar coagulation, hemostasis will be performed using bipolar tweezers as few times as possible, just to control any considerable bleeding, at 30 W; the number of coagulated points will be recorded, and the duration of the procedure at each bleeding point will measured. These parameters will help elucidate possible flaws in previous studies, in which assessments were subjective, without specification of the duration of the coagulation in each point or the number of coagulated points.

In the group allocated to receive hemostasis by means of laparoscopic surgery, bipolar coagulation will not be performed, and the procedure will involve simple intraovarian sutures 1 or 2 knots with 2-0 Vicryl; the number of sutures will be counted.

In the group allocated to receive hemostasis by means of hemostatic matrix, bipolar coagulation will not be performed, and the sealant will be applied on the ovarian wound surface.

Procedures for data collection

Data collection instrument. The data will be recorded on standardized forms containing closed-ended questions pre-encoded for entry into the computer.

The information corresponding to categorical variables will be pre-encoded. Continuous variables will be expressed in the corresponding numerical values; only at the time of analysis will some be categorized.

The forms will be duly stored in specific folders before and after typing and analysis. This task will be under the responsibility of the investigator, who will complete the forms at various time points.

Data collection. The data will be collected by the investigator and a collaborator, who is a student from the Institutional Program of Undergraduate Research Scholarships. The collaborator will apply the checklist to candidates according to the eligibility criteria. Next, the study protocol will be applied, and the forms will be completed to record all necessary information.

Once completed, the forms will be rigorously reviewed by the investigator to check the collected information against that in the medical records. The time-points for data collection, adequate form completion and review will comply with those indicated in the schedule.

Data analysis. Statistical analysis will be performed by the investigator, her supervisors and a statistician using Excel software and the statistical software SPSS for Windows, version 19.0.0. Originally, SPSS was the acronym for Statistical Package for the Social Sciences, but at the present time, it is a part of the software name IBM SPSS®, without indication of any particular meaning.

Numerical variables will be compared by means of one-way analysis of variance ANOVA or the Kruskal-Wallis tests according to the normality or non-normality of the distribution. The chi-square or Fisher's tests will be used for categorical variables.

DISCUSSION

The reduction of ovarian function among patients with endometrioma is still a subject of study, and its cause requires further elucidation. Some authors consider that the presence of endometrioma itself accounts for the impairment of ovarian function. According to other authors, the factor associated with such impairment is the hemostatic method used following stripping of the endometrioma capsule, as some studies indicate that bipolar coagulation causes greater ovarian damage. However, no study has objectively assessed either the number of points requiring coagulation or the duration of coagulation; furthermore, the energy used is not standardized among studies. The present study intends to assess the ovarian function of patients with endometrioma subjected to laparoscopic surgical treatment, comparing different hemostatic techniques (bipolar coagulation versus suture versus hemostatic matrix) with objective assessments of bipolar coagulation to avoid bias. Thus, the investigators expect to contribute data likely to dispel doubts on the subject.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Regular menstrual cycle (21 to 35 days).
* Unilateral ovarian cyst suggestive of endometrioma.
* Endometrioma and indication of laparoscopic surgery for cyst removal due to pelvic pain, infertility or cyst persistence.

Exclusion Criteria:

* Previous ovarian surgery.
* Endocrine dysfunction (diabetes, thyroid disorders, hyperprolactinemia, adrenal disease, polycystic ovary syndrome).
* Use of hormones in the past 3 months.
* Suspected ovarian malignant tumor requiring oophorectomy.
* History of chemotherapy or radiotherapy.
* Coagulation disorders.
* Pregnancy.
* Autoimmune disease.

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
AMH | Before surgery
  Antimullerian hormone levels
AMH | 1month after the surgery
  Antimullerian hormone levels
AMH | 3 months after the surgery
  Antimullerian hormone levels
AMH | 6 months after the surgery
  Antimullerian hormone levels

SECONDARY OUTCOMES:
AFC | Before surgery
  Ultrasound antral follicle counts
AFC | 1month after the procedure
  Ultrasound antral follicle counts
AFC | 3 months after the procedure
  Ultrasound antral follicle counts
AFC | 6 months after the procedure
  Ultrasound antral follicle counts

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Araujo, M.D., Principal Investigator — Faculdade de Ciências Médicas da Santa Casa de São Paulo; Universidade Federal da Paraíba
Locations (1):
- Universidade Federal da Paraiba, João Pessoa, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Araujo RSDC, Maia SB, Baracat CMF, Fernandes CQBA, Ribeiro HSAA, Ribeiro PAAG. Ovarian function following use of various hemostatic techniques during treatment for unilateral endometrioma: A randomized controlled trial. Int J Gynaecol Obstet. 2022 Jun;157(3):549-556. doi: 10.1002/ijgo.13912. Epub 2021 Sep 21. PMID 34478564